CLINICAL TRIAL: NCT02790346
Title: Interest of Talonavicular Arthrodesis on Walking Speed at Brain Lesion Patients Who Benefit of a Surgical Treatment of Ankle and Varus Foot : Randomized Study
Brief Title: Talonavicular Arthrodesis and Surgical Treatment of Ankle and Varus Foot
Acronym: talobot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9547
Record Dates: First submitted 2016-05-17; First posted 2016-06-03 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Orthopedic Equine Varus Deformity
Keywords: hemiparesis; deformity of the foot and ankle
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arthrodesis talonavicular (Experimental): arthrodesis talonavicular in addition to tendon gestures
  Interventions: Procedure: arthrodesis talonavicular; Procedure: tendon gestures
- tendon gestures (Active Comparator): tendon gestures only
  Interventions: Procedure: tendon gestures

INTERVENTIONS:
Procedure: arthrodesis talonavicular
  Arms: arthrodesis talonavicular
Procedure: tendon gestures

SUMMARY:
This study should refine our surgical indications and to establish a decision tree of medical and surgical treatment of this common and troublesome strain functionally which is equino-varus.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis secondary to a lesion of the central nervous system, regardless of the etiology dated within 6 months
* Orthopedic equine-varus deformity of the foot and ankle requiring surgery
* Patient able to move by walking preoperatively at least 2 meters with or without technical assistance or may earn postoperative walking ability

Exclusion Criteria:

* History of foot surgery the side to be operated
* Significant deformation set foot and ankle (requiring treatment with triple arthrodesis)
* Bilateral surgery
* Progressive neurological disease
* Dystonic movements or movement disorders
* Realization of a botulinum toxin injection in the 6 months preceding gesture
* Important cognitive impairment

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
walking speed at one year | 12 months after surgery intervention

SECONDARY OUTCOMES:
walking speed at 3 and 6 months | 3 months and 6 months after surgery intervention

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Lapeyronie, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No